CLINICAL TRIAL: NCT02093078
Title: Cognitive Aids With Roles Defined (CARD) for Obstetrical Crises: A Multisite Cohort Study
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20120926-01H
Record Dates: First submitted 2014-02-07; First posted 2014-03-20 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Obstetrical Emergency Situations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CARD: Intervention: CARD
  This group will be introduced to the CARD protocol which focuses on clarification of individual roles and distribution of tasks. It relies on large identification cards specially designed for each team member's profession and role. Each card worn by a team member identifies the specific tasks associated with that individual's role. CARD enables the team leader and other team members to quickly recognize everyone's role at the code, and each team member can commence their assigned tasks without delay.
  Interventions: Behavioral: CARD
- Control Arm

INTERVENTIONS:
Behavioral: CARD — Intervention: CARD
  This group will be introduced to the CARD protocol which focuses on clarification of individual roles and distribution of tasks. It relies on large identification cards specially designed for each team member's profession and role. Each card worn by a team member identifies the specific tasks associated with that individual's role. CARD enables the team leader and other team members to quickly recognize everyone's role at the code, and each team member can commence their assigned tasks without delay.
  Groups: CARD

SUMMARY:
Crisis resource management represents the set of non technical skills, such as communication, leadership, delegation, and prioritization, that allow effective teamwork for optimal patient care during an urgent and critical situation. The Cognitive Aids with Roles Defined (CARD) is a new concept of cognitive aid addressing the well-documented issue of teamwork in crisis management. It relies on large identification cards specially designed for each team members profession and role. During a life threatening clinical situation, the CARD protocol focuses on clarification of individual roles and distribution of tasks for crisis management rather than creating an additional algorithm identifying either a list of actions to be taken or the dose of a medication. This study aims to evaluate the clinical impact of introducing the CARD protocol in obstetrical emergency situations ("code 333") in clinical practice at The Ottawa Hospital.

Hypothesis: CARD protocol will: (i) decrease the total time taken to deliver the baby, and (ii) improve clinical outcome for the mother and baby compared to traditional management without the CARD protocol.

DETAILED DESCRIPTION:
The CARD protocol offers an innovative yet simple solution to the barriers in crisis management that the literature has already identified. The study is part of a research program investigating strategies to improve crisis management. After completing several simulation studies on cognitive aids, crisis management debriefing, and a pilot CARD study, the investigators aim to explore and investigate the impact of an intervention on patient care.

The concept of a self-organizing team with explicitly defined roles may enhance patient safety. The CARD approach to crisis management is relevant to a broad number of situations, disciplines, and professions. The CARD protocol is easily exportable to any critical situation including intra-hospital arrest, trauma, or critical care patients. The concept of a self-organizing team with defined roles may ultimately enhance patient safety.

The investigators anticipate that their proposal will challenge the traditional way of thinking about cognitive aid, and may advance the theory in the two fields of cognitive aid and team work for crisis management.

The CARD cards with their associated roles and list of tasks will be specifically designed for code 333. In the 'baseline' phase, a research assistant will review Birthing Unit records daily to determine if a code 333 had been called in the preceding 24 hours. Outcome measures will be collected to establish baseline team performance. In order to account for the 'team training effect' and identify the 'CARD effect', both groups will receive didactic and simulation crisis management teaching, but training at the "case site" will include CARD teaching while the contemporaneous "control site" will receive team training without CARD. After the training period at both sites, CARD will be implemented at the "case sight" for code 333s while the "control site" will continue without CARD. Maternal and neonatal outcomes as well as team performance (times to delivery) will continue to be prospectively collected throughout.

ELIGIBILITY:
Inclusion Criteria:

* must hold a staff position at The Ottawa Hospital (Civic or General campus) in one of the following positions:

  1. registered nurses (RN)
  2. operating room attendant
  3. respiratory therapist (RT)
  4. assisting anesthesia
  5. RT assisting neonatal
  6. neonatal RNs

     Exclusion Criteria:
* not a staff member at The Ottawa Hospital (Civic or General campus)
* holding a position that is different from any of the following: registered nurse, operating room attendant, respiratory therapist, assisting anesthesia, RT assisting neonatal, neonatal RN
* investigators involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twelve obstetrical unit teams (4 registered nurses (RN), 1 operating room attendant, 1 respiratory therapist (RT) assisting anesthesia, 1 RT assisting neonatal, 2 neonatal RNs) will be recruited for the study
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Total Time to Delivery After a Code 333 | from the time of calling in a code 333 to the time of birth (up to 1 day).
  The primary outcome measure is the exact time from when the code 333 is called, to the time of delivery (up to 1 day).

SECONDARY OUTCOMES:
standard clinical outcomes on patient charts | participants will be followed from when the code 333 was called until hospital discharge or mortality, whichever comes first (up to 3 years).
  The clinical outcomes on patient charts include:
  Baby's status:
  1. Apgar score, at 1 and 5 minutes
  2. Arterial potential hydrogen (pH) of the cord at birth
  3. Unplanned admission to intensive care for the baby
  4. Infant status at 1 hour of age
  5. Length of stay of the baby in hospital
  6. Mortality
  Mother clinical outcomes:
  1. Unplanned admission to ICU for the mother
  2. Length of stay of the mother in hospital
  3. Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada